CLINICAL TRIAL: NCT06738550
Title: Effect of Agave Inulin on Constipation and Quality of Life in Peritoneal Dialysis Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: NIN Institute (Industry)
Responsible Party: Principal Investigator, Ari Cisneros-Hernández, Principal Investigator, Centro Medico Issemym
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NI0002/24
Record Dates: First submitted 2024-09-23; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Constipation; Peritoneal Dialysis (PD); CKD; Quality of Life (QOL)
Keywords: CKD; Peritoneal Dialysis (PD); Constipation; Quality of life (QOL); Gastrointestinal symtoms
MeSH Terms: conditions — Constipation | interventions — Inulin; Lactulose

STUDY DESIGN:
Intervention Model Description: control group with lactulose syrup 10 ml every 8 hours and nutritional intervetion intervention group with agave inulin 9 gr per day and nutritional intervetion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inulina (Experimental): In the patients of the experimental group, the nutritional intervention is personalized, agave inulin supplementation is provided 9 gr per day, A 6-month follow-up is provided
  Interventions: Dietary Supplement: inulin
- Lactulosa (Placebo Comparator): In the patients of the control group, the nutritional intervention is personalized, A 6-month follow-up is provided and taken syrup lactulose 10 ml every 8 hours
  Interventions: Drug: Lactulose oral solution

INTERVENTIONS:
Dietary Supplement: inulin — In the patients of the experimental group, the nutritional intervention is personalized, agave inulin supplementation is provided 9 gr per day, A 6-month follow-up is provided
  Other Names: Inulin prebiotic
  Arms: Inulina
Drug: Lactulose oral solution — In the patients of the experimental group, the nutritional intervention is personalized, A 6-month follow-up is provided and taken syrup lactulose 10 ml every 8 hours
  Arms: Lactulosa

SUMMARY:
This is a randomized controlled clinical study realized in the nephrology service of the Centro Medico ISSEMyM hospital in Metepec, State of Mexico, including new patients on Peritoneal Dialysis (PD) over 18 years of age with constipation criteria, the Bristol scale and Rome IV Criteria were used, with a 6-month follow-up with a personalized diet plan, intervention group supplementation with agave Tequiliana blue variety inulin with an initial dose of 9 grams per day, the control gruop recived lactulosa. Data were obtained from the clinical history comorbidities present in the patients, anthropometric data such as weight, % of fat, % of body water, Fat Free Mass (FFM) obtained using a TANITA scale model BC-533; skin folds were obtained using a slim Guide plicometer, dietary data such as energy intake (kcal), protein intake, fluid intake, were estimated using a 24 hr reminder. A questionnaire was also applied to measure gastrointestinal symptoms and their evolution with the intervention, in addition to the KDQOL-SF to evaluate the quality of life of the patients.

DETAILED DESCRIPTION:
Constipation affects a large part of the population with Chronic Kidney Disease (CKD), and in Peritoneal Dialysis (PD) it is the most common symptom derived from multiple factors, including dietary restrictions causing insufficient fiber intake, water restriction, drug consumption and the change in the intestinal microbiota derived from uremic toxins during this stage, leading to a poor quality of life in the patient and consequently an alteration in the patient's nutritional status. In turn, constipation has become a risk factor in the development of cardiovascular diseases, of which patients with CKD have a higher incidence. This research aims to determine the effects of agave inulin supplementation on constipation and quality of life in peritoneal dialysis patients in order to establish a strategy to support patient treatment and improve uremic syndrome.

Lactulose syrup is usually used to prevent and treat constipation in doses from 10 ml every 8 hours.

The present research aims to determine the effects that agave inulin supplementation may have on constipation and quality of life in peritoneal dialysis patients, and to establish a strategy to support the patient's treatment and improve uremic syndrome.

Stage 1 Patients will be selected by the peritoneal dialysis team to identify the patients who start RRT, once identified, they will be referred to the nutrition office, where an initial evaluation of the patient will be made and if they meet the inclusion criteria, the informed consent will be explained and if they accept, they will be randomly assigned to the group they are assigned to. The laboratories requested to the patients are the same as those routinely requested by the treating physician. The characteristics of the nutritional intervention are detailed below. The characteristics of the first visit are detailed below.

Visit 1:

1. Evaluation of selection/inclusion criteria
2. Assessment in medical consultation
3. Signing of consent form.
4. Initial evaluation (File with: clinical, anthropometric, biochemical, dietary data).
5. Constipation evaluation with Bristol scale
6. Evaluation of quality of life with KDQOL-SF questionnaire.
7. Delivery of food plan and nutritional recommendations
8. Indication and delivery of the supplement according to the group.
9. Indicate that unfinished product should be returned.
10. Request for laboratory tests (routine tests that the nephrologist requests consultation after consultation).
11. Appointment every 30 days for delivery of supplement and adherence evaluation.

Stage 2 In the second stage, patients are followed month by month for medical and nutritional evaluation, evaluating anthropometry, biochemistry, clinical signs, patient's diet, therapeutic adherence to supplementation, evaluation of gastrointestinal symptoms and constipation, and evaluation of quality of life. The corresponding data are recorded in a database. The characteristics of the visit are detailed below.

Visit 2, 3, 4 and 5:

1. Intermediate medical evaluation
2. Intermediate evaluation (File with: clinical, anthropometric, biochemical, dietary data, adherence evaluation).
3. Constipation evaluation with Bristol scale and roma criteria.
4. Supplement delivery
5. Request for laboratory tests (routine tests requested by the nephrologist consultation after consultation).
6. Appointment every 30 days.

Stage 3 In this stage the supplementation is suspended, a medical and nutritional evaluation is made evaluating anthropometry, biochemistry, clinical signs, patient's diet, therapeutic adherence to supplementation, evaluation of gastrointestinal symptoms and constipation and evaluation of quality of life. The corresponding data are recorded in a database. The characteristics of the visit are detailed below.

Visit 6: discontinue supplementation.

1. Final evaluation (clinical record with anthropometric, clinical, biochemical and dietary data, evaluation of therapeutic adherence).
2. Evaluation of constipation with Bristol scale and roma criteria.
3. Request for laboratory tests (routine tests that the nephrologist requests consultation after consultation).
4. Appointment after 30 days. In this last stage, the patient will be seen again after one month to evaluate the post-supplementation period.

In this last stage, the patient will be seen again after one month to evaluate the post-supplementation period.

Visit 7:

1. Post-intervention period evaluation (file with: clinical, anthropometric, biochemical, dietary data).
2. Evaluation of constipation with Bristol scale and roma criteria.
3. Evaluation of quality of life with KDQOL-SF questionnaire.

Characteristics of the nutritional intervention:

In the nutritional intervention, the patient's family medical history, clinical indicators such as T/A, signs of nutritional deficiency such as dehydration, muscle and fat depletion, edema and gastrointestinal symptoms and degree of constipation will be evaluated by clinical history.

Biochemical indicators are tests that are commonly requested in nephrology follow-up consultations, will be evaluated.

For the evaluation of anthropometric indicators, body composition will be evaluated by means of anthropometry (plyometry and circumferences) and a Tanita scale, identifying the patient's fat and muscle compartment; in the dietary evaluation, the intake of energy, carbohydrates, lipids and proteins will be evaluated by means of a 24-hour reminder. With the above, a nutritional diagnosis is made and a dietary plan for the patient that includes: general recommendations, explanation of portions, explanation of the food for renal disease and a menu with food options that the patient can follow and exchange with the list of foods provided.

Ethical considerations. Requesting their signature for consent. Human research guidelines will be respected according to "good clinical practice". The protocol will be submitted to the Bioethics Committee of the Centro Medico ISSEMyM, Metepec, Edo. México. Care will be taken to respect the recommendations of the Helsinki Declaration in its last correction made during the 64th Annual Assembly organized by the World Medical Association (2013).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Beginning of peritoneal dialysis in the last month
* Constipation
* Medical follow-up by nephrology every month
* Without Irritable Bowel Syndrome
* No frailty criteria

Exclusion Criteria:

* Patients who don't to take the supplement
* Patients with diarrhea
* Patients with a diagnosed intestinal disorder
* Allergic to any ingredient of the supplement.
* Previous probiotic and/or prebiotic supplementation in the last month
* Diagnosis of comorbidities such as cancer, decompensated heart failure, decompensated pulmonary disease, decompensated liver disease, HIV, infection present within the last 3 months (chronic and/or acute), stroke and malabsorption syndrome.
* Hospitalizations within the last month for peritonitis
* Pregnant women
* Patients with psychiatric illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Constipation | Baseline intervetion and 6 months
  Change stool consistency as assessed by the Bristol scale
  1 and 2 is Cosntipacion 3 and 4 is Normal 5, 6 and 7 is diarrhea
Gastrointestinal symptoms | Baseline intervention and 6 months
  Changing the intensity of gastrointestinal symptoms caused by CKD and constipation as assessed with the PAC-SYM QUESTIONNAIRE
  Designed to assess the patient's experience of constipation over two weeks by measuring symptoms and symptom severity. It is a self-reported questionnaire consisting of 12 symptoms divided into three domains: abdominal, rectal and stool, with responses rated on a 5-point Likert scale.
  Scoring The PAC-SYM is a tool that can be used to understand the severity of your patient's constipation and help you identify key symptom areas. A total PAC-SYM score ranges from 0 to 48 with a low score indicating fewer symptoms and of lower severity.
  Absence of symptom = 0 Mild = 1 Moderate = 2 Severe = 3 Very severe = 4

SECONDARY OUTCOMES:
Dietary intake (kcal/kg/day) | baseline intervention and 6 months
  Changes in dietary caloric intake of patients at baseline and month 6

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Medico ISSEMyM, Toluca, Metepec, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: No